CLINICAL TRIAL: NCT00457678
Title: A Multicenter, Randomized, Single-Masked Comparison of Lucentis™ Monotherapy With Triple Therapy of Reduced Fluence Visudyne-Lucentis-Dexamethasone (V-L-D) in Patients With CNV Secondary to AMD as Second Line Therapy After Lucentis Monotherapy
Brief Title: Second Line Therapy to Treat Age-related Macular Degeneration (AMD) for Patients Not Responding Well to Lucentis Therapy by Itself
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Site did not enroll any patients to the study.
Sponsor: Vitreous -Retina- Macula Consultants of New York (Other)
Collaborators: QLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAPER
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Age Related Macular Degeneration
Keywords: Vision loss; Retina; VEG-F; Fovea; AMD
MeSH Terms: conditions — Macular Degeneration; Vision Disorders | interventions — Verteporfin; Ranibizumab; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients with
  AMD will be randomly assigned to one of 2 treatments:
  * Continuation of previous Lucentis monotherapy (50 patients)
  * V-L-D triple therapy with half fluence (300 mW/cm2 for 83 seconds) Visudyne followed within 2 hours by intravitreal Lucentis 0.5 mg (first injection) and intravitreal dexamethasone 0.5 mg (second injection) (50 patients)
Who Masked: Participant

INTERVENTIONS:
Drug: Visudyne
Drug: Lucentis
Drug: Dexamethasone

SUMMARY:
The purpose of this study is to demonstrate that Visudyne-Lucentis-dexamethasone (V-L-D) triple therapy will give similar efficacy and safety results as Lucentis monotherapy.

DETAILED DESCRIPTION:
Study Design:

Patients who have received 2-6 previous treatments with Lucentis monotherapy and who have exudative activity associated with the choroidal neovascularization (CNV) lesion, as confirmed by fluorescein angiography (FA) or optical coherence tomography (OCT), will be eligible. Patients will be randomly assigned at 4-8 weeks after the previous Lucentis treatment to either

1. continuation of Lucentis monotherapy
2. triple therapy with half fluence Visudyne (300 mW/cm2 for 83 seconds) followed within 2 hours by intravitreal Lucentis 0.5 mg (first injection) and then dexamethasone 0.5 mg (second injection) (V-L-D).

Both groups will receive treatment at baseline and then as needed (PRN), according to retreatment criteria, with monthly assessments thereafter for 12 months. In the triple therapy group, patients may only be retreated with the V-L-D combination at intervals of no less than 3 months; if retreatment is needed 1 or 2 months after a previous V-L-D treatment, the patient will receive a Lucentis injection at that visit; however, if retreatment is needed and the previous V-L-D treatment was at least 3 months prior, then V-L-D treatment is mandatory. OCT, visual acuity (VA) testing, and possibly FA will be conducted at each assessment visit to define the need for retreatment.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with subfoveal CNV due to AMD who, after 2-6 previous treatments with Lucentis monotherapy, continue to have exudative activity associated with the CNV lesion 4-8 weeks after the last treatment. Exudative activity is defined as one or more of:

  * CNV leakage confirmed by FA
  * New hemorrhage associated with the CNV lesion
  * Subretinal fluid or cystoid macular edema by OCT showing retinal thickness ≥ 230 μm
* All lesion composition types with a lesion greatest linear dimension (GLD) ≤ 5400 microns (approximately ≤ 9 disc areas [DA])
* Best corrected ETDRS VA score of 25-73 letters (approximate Snellen equivalent of 20/40-20/320)

Main Exclusion Criteria:

* Subfoveal geographic atrophy or subfoveal fibrosis in the study eye
* Intraocular surgery within 3 months of enrollment
* Inability to attend the protocol-required visits
* Known allergies or hypersensitivity to any of the study treatments

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01 (Estimated); Primary Completion 2007-12-04 (Actual); Study Completion 2007-12-04 (Actual)